CLINICAL TRIAL: NCT05630222
Title: Evaluation of Effect of Intravenous Morphine vs Intravenous Ibuprofen and Acetaminophen vs Intravenous Ibuprofen on Pain Relief in Patients With Closed Extremity Fracture Admitted in Alzahra and Ayatollah Kashani Hospitals in 2022
Brief Title: Evaluation of Effect of Intravenous Morphine vs Intravenous Ibuprofen and Acetaminophen vs Intravenous Ibuprofen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Associate Professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3401308
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Multiple Trauma; Acute Pain Due to Trauma
MeSH Terms: conditions — Multiple Trauma | interventions — Ibuprofen; Morphine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ibuprofen (Active Comparator): Ibuprofen 800 mg IV infusion over 20 min.
  Interventions: Drug: Ibuprofen 800 mg
- Morphine (Active Comparator): Morphine Sulfate 0.1 mg/kg IV
  Interventions: Drug: Morphine Sulfate
- Ibuprofen plus Acetaminophen (Active Comparator): Ibuprofen 400 mg plus Acetaminophen 1000 mg IV infusion over 20 min.
  Interventions: Drug: Ibuprofen 400 mg plus Acetaminophen 1000 mg

INTERVENTIONS:
Drug: Ibuprofen 800 mg — Ibuprofen from Caspian Taamin Company
  Arms: Ibuprofen
Drug: Morphine Sulfate — Morphine Sulfate from Darupakhsh Company
  Arms: Morphine
Drug: Ibuprofen 400 mg plus Acetaminophen 1000 mg — Both from Caspian Taamin Company
  Arms: Ibuprofen plus Acetaminophen

SUMMARY:
Pain is an inseparable symptom of fractures and is the most important and common symptom that brings patients to medical centers; Therefore, paying attention to pain and its control is very important in the examination and treatment of fractures, and painkillers are usually needed for effective pain control. About 70-90% of the patients who go to the emergency room due to injuries have organ injuries. Among these patients, those who suffer from fractures endure severe pain, and since only 10% of patients have open fractures, the pain management of patients with closed fractures is particularly important. Various medicinal compounds have been used so far to control the pain of fractured patients, including opioid compounds such as morphine, non-steroidal anti-inflammatory drugs such as ibuprofen and acetaminophen. Opioids are the main drug class for pain control in fractures, but since they have significant side effects, various studies have been conducted in the field of comparing the anti-inflammatory effect of different drugs in fractures, and the effect of various combinations compared to opioids has been investigated. Non-steroidal anti-inflammatories are always considered as an alternative to opioids and acetaminophen has also been considered to reduce the dosage of opioids, so in this study the effect of three combinations of intravenous morphine and ibuprofen plus intravenous acetaminophen and intravenous ibuprofen on pain levels in patients with a closed limb fracture will be investigated.

This study is a blind randomized clinical trial, which investigates and compares the effect of intravenous morphine (Daropakhsh Company) with intravenous ibuprofen (Caspian Taamin Company) and intravenous acetaminophen (Caspian Taamin Company) with intravenous ibuprofen (Caspian Taamin Company) in reducing the pain of patients with closed limb fractures. The population investigated in this study will include all patients referred to the emergency room of Al-Zahra and Ayatollah Kashani educational centers in Isfahan city in 2022-2023.

DETAILED DESCRIPTION:
The study subjects are classified into 3 groups by computerized random allocation method, the first group will receive 0.1 mg/kg of intravenous morphine (Daropakhsh company) and the second group will take 400 mg of intravenous ibuprofen (Caspian Taamin company) plus 1 gram of intravenous acetaminophen (Caspian company). Tamin) and the third group receives 800 mg of intravenous ibuprofen (Caspian Taamin Company).This study is a blind randomized clinical trial, which investigates and compares the effect of intravenous morphine with intravenous ibuprofen and intravenous acetaminophen with intravenous ibuprofen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing a closed fracture of any of the bones of the body by an emergency medicine specialist
* Informed consent of the patient or his family to participate in the study
* Age 18 to 55 years
* Pain score of higher than or equal to 6 on the VAS scale
* Informed consent of the patient or family during the study
* No history of liver or kidney failure
* No history of gastrointestinal bleeding
* No history of heart failure
* No history of allergy to study drugs
* Absence of addiction (the patient is asked)
* Not decreased level of consciousness
* Lack of evidence of increased intra-cerebral pressure
* Not having an open fracture
* Absence of breathing disorders and respiratory problems
* No history of asthma
* Lack of history of frequent use of painkillers
* Not receiving any form of pain killer in the last few hours

Exclusion Criteria:

* Occurrence of any type of drug reaction or unusual complication during the study period
* Simultaneous Head trauma
* Simultaneous damage of nerves and blood vessels
* Multiple fractures
* Fracture other than limb
* Evidence of increased intra-cerebral pressure
* Decreased level of consciousness
* Breathing disorders and respiratory problems

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue score (VAS) | Change from baseline at 60 minutes
  a scale for measuring the extent of pain relief

SECONDARY OUTCOMES:
HR | Change from baseline at 60 minutes
  Heart rate
RR | Change from baseline at 60 minutes
  Respiratory rate
SpO2 | Change from baseline at 60 minut
  Blood oxygen saturation
BP | Change from baseline at 60 minut
  Blood Pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahra University Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
It will be possible to share data if requeste
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Nasr Isfahani M, Etesami H, Ahmadi O, Masoumi B. Comparing the efficacy of intravenous morphine versus ibuprofen or the combination of ibuprofen and acetaminophen in patients with closed limb fractures: a randomized clinical trial. BMC Emerg Med. 2024 Jan 25;24(1):15. doi: 10.1186/s12873-024-00933-y. PMID 38273252